CLINICAL TRIAL: NCT05977400
Title: NICU Antibiotics and Outcomes Follow-Up Study
Brief Title: NICU Antibiotics and Outcomes (NANO) Follow-up Study
Acronym: NANO-FU
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Collaborators: University of Pittsburgh (Other); Morgan Stanley Children's Hospital (Other); University of Louisville (Other); Sharp Mary Birch Hospital for Women & Newborns (Other); Children's Hospital of Philadelphia (Other); Jefferson Medical College of Thomas Jefferson University (Other); University of South Florida (Other); Westchester Medical Center (Other); Yale University (Other); The University of Texas Health Science Center at San Antonio (Other); Penn State University (Other); State University of New York - Downstate Medical Center (Other); Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Anup Katheria, M.D., PI, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NANO Follow-Up
Record Dates: First submitted 2021-05-24; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Premature Birth; Antibiotics; Neurodevelopment
MeSH Terms: conditions — Premature Birth | interventions — Ampicillin; Gentamicins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Very preterm infants that receive empiric antibiotic treatment in the first 48 hours of life (Active Comparator): Neonates in this group will have been enrolled and randomized into the NANO trial and received a blinded 48 hour course of empiric antibiotic treatment.
  Interventions: Drug: Ampicillin; Drug: Gentamicin
- Very preterm infants that do not receive empiric antibiotic treatment in the first 48 hours of life (Placebo Comparator): Neonates in this group will have been enrolled and randomized into the NANO trial and received a blinded 48 hour course of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ampicillin — Intravenous Ampicillin
  Arms: Very preterm infants that receive empiric antibiotic treatment in the first 48 hours of life
Drug: Gentamicin — Intravenous Gentamicin
  Arms: Very preterm infants that receive empiric antibiotic treatment in the first 48 hours of life
Drug: Placebo — Intravenous Normal Saline
  Arms: Very preterm infants that do not receive empiric antibiotic treatment in the first 48 hours of life

SUMMARY:
The NANO follow-up study is designed to determine whether a simple, cost-effective intervention- withholding antibiotics at birth- reduces clinically relevant outcomes such as behavioral and neurological impairment at 2 years of age. This study will be the largest study evaluating the effects of early antibiotics in children with comprehensive measures of neurodevelopment linked to genomic variants and microbiota interactions.

DETAILED DESCRIPTION:
The multidisciplinary team launched the NANO (NICU Antibiotics and Outcomes) Trial to study the longstanding clinical practice of empirically administering intravenous antibiotics to very preterm infants. The NANO trial is an 802-patient,13-site randomized blinded controlled trial (R01HD09757801) discerning whether administration of antibiotics within the first three days of life increases the incidence of short-term, life-threatening complications among very preterm infants.

The proposed NANO follow-up study will build upon the parent NANO trial to determine whether avoiding antibiotics in very preterm infants - a simple, cost-effective intervention - improves neurodevelopmental and behavioral outcomes during the toddler years. Evaluation of children enrolled in the proposed NANO follow-up study will include serial comprehensive, standardized assessments of motor, cognitive, behavioral and adaptive outcomes. To support retention and provide an important early assessment, a first virtual visit at 1 year of age will include the Hammersmith Infant Neurologic Exam (HINE) and the Developmental Assessment of Young Children, Second Edition (DAYC-2). A second comprehensive follow-up visit in person at 2 years will include the Bayley Scales of Infant Development 4th ed., Gross Motor Function Classification System, Child Behavior Checklist for ages 1.5-5, and the Modified Checklist for Autism in Toddlers, Revised, with Follow-up.

In the NANO follow-up trial, outcomes will be assessed using the Desirability of outcome ranking (DOOR), an innovative, patient-centered statistical approach used in clinical trials to evaluate the global benefits and risks of an intervention. The ordinal neonatal follow-up endpoint composite scale, to be named neoDOOR, will be developed by both clinicians and families. Stakeholder meetings will develop consensus rankings of individual and composite outcomes of different severities reported by the above developmental assessments. Neonatal biospecimens collected during the parent NANO trial will allow for additional exploratory analyses evaluating interactions among genetics, environment, and microbiota with antibiotic exposure and long-term outcomes. Through these assessments and evaluation, the investigators will provide substantial evidence for the use (or non-use) of early antibiotics for very preterm infants at birth.

ELIGIBILITY:
Inclusion Criteria: Families that have agreed to participate and are enrolled in the parent NANO trial will be eligible for the NANO follow-up study. There will be no exclusions for eligible children entering the follow-up study.

Parent NANO trial Criteria:

I. Inclusion criteria: We will enroll newborn infants with gestational age of 23.0-30.6 weeks born to mothers 18 years or older at participating study sites. Only inborn infants at participating study sites will be eligible.

II. Exclusion criteria:

1. Infants at low risk for early onset sepsis-Infants born for maternal indications via caesarean section with rupture of membranes within 6 hours, without attempts to induce labor, and without concern for maternal infection
2. Infants at high risk for early onset sepsis- Infants born to mothers with intrapartum fever (> 38ºC) or clinical diagnosis of chorioamnionitis (suspected or definite), infants born to mothers with proven Group B Streptococcus colonization or indication for intrapartum antibiotic prophylaxis that did not receive adequate antibiotic treatment according to specialty specific guidelines, (i.e., penicillin, ampicillin, cefazolin), infant born to mother with previous infant with GBS disease/infection
3. Infants with respiratory insufficiency requiring invasive mechanical ventilation and fraction of inspired oxygen> 0.40 or non-invasive ventilation and fraction of inspired oxygen > 0.60 at time of randomization
4. Infants with ongoing hemodynamic instability requiring vasopressors or more than one fluid bolus at time of randomization
5. Clinician concern for sepsis due to physical exam findings or clinical history of mother or infant
6. Major congenital anomalies
7. Infants not anticipated to survive beyond 72 hours
8. Infants who have received antibiotics prior to randomization.

Ages: 23 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 802 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Rate of neurodevelopmental impairment or Death | 24 months corrected gestational age
  The first primary outcome will be a composite of newborn or childhood death OR one of following: cognitive or motor composite scores <80 on the Bayley-4, Gross Motor Function Classification Score score ≥2, bilateral blindness, severe functional hearing impairment. The incidence of the composite outcome will be compared between the placebo and early antibiotic groups.
DOOR probability Distribution | 24 months corrected gestational age
  The second primary outcome will be a comparison of the DOOR probability of more desirable outcomes at 2 years using a novel ordinal endpoint scale developed during the trial. Outcomes to be included in the rank are as follows: death, cognitive/language/motor composite scores<80 on the Bayley-4, Gross Motor Function Classification Score ≥2, bilateral blindness, severe functional hearing impairment, Child Behavior Checklist (CBCL) scores >70, autism risk scores (MCHAT R/F) of ≥2, and medical measures, such as need for oxygen support. The distribution of the finalized neoDOOR will be compared between the placebo and empiric antibiotic groups.

CONTACTS AND LOCATIONS:
Overall Officials: Anup Katheria, MD, Principal Investigator — Sharp HealthCare
Locations (15):
- United States (14):
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California
  - Yale University, New Haven, Connecticut
  - University of South Florida, Tampa, Florida
  - University of Louisville, Louisville, Kentucky
  - State University of New York Downstate, Brooklyn, New York
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - Westchester Medical Center, Valhalla, New York
  - The Pennsylvania State University, Hershey, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Jefferson Medical College of Thomas Jefferson University, Philadelphia, Pennsylvania
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - The University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Sinai Health System, Toronto, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available per NICHD requirements (National Institute of Child Health and Human Development).
Supporting Information: SAP
Time Frame: 2 years after primary publication
Access Criteria: An archived dataset with documentation will be made available for additional uses by outside investigators, in collaboration with the study investigators. We will work with NICHD program staff to develop a broad data sharing plan over time.